CLINICAL TRIAL: NCT00663117
Title: The Effects of Naltrexone in Active Crohn's Disease
Brief Title: The Effects of Naltrexone on Active Crohn's Disease
Acronym: LDN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Broad Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK073614 l; 1R03DK073614 (NIH); IBD-0180R (Other Grant/Funding Number: Broad Medical Research Program)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2013-05

CONDITIONS: Inflammation; Crohn's Disease
Keywords: naltrexone; LDN; IBD; Inflammatory bowel disease
MeSH Terms: conditions — Inflammation; Crohn Disease; Inflammatory Bowel Diseases | interventions — Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo, Sugar pill (Placebo Comparator): placebo for 3 months blinded then followed by an open-labelled study and all are treated with naltrexone 4.5 mg for 3 additional months
  Interventions: Drug: Naltrexone-HCl; Drug: Placebo
- Naltrexone-HCl (Active Comparator): Subjects are treated in a blinded fashion for 3 months with naltrexone 4.5 mg po for active Crohn's disease followed an open-labelled study where naltrexone is given an additional 3 months at 4.5 mg po; hence the total treatment interval in this arm is 6 months. The response to the intervention administered is measured in the activity index and mucosal healing by colonoscopy.
  Interventions: Drug: Naltrexone-HCl

INTERVENTIONS:
Drug: Naltrexone-HCl — naltrexone 4.5 mg
  Other Names: LDN; Revia
Drug: Placebo — Placebo
  Other Names: sugar pill
  Arms: Placebo, Sugar pill

SUMMARY:
It is hypothesized that the opioid antagonist naltrexone will improve inflammation of the bowel and quality of life in subjects with active Crohn's disease compared to placebo. In order to test this hypothesis the following specific aims are proposed:

1. Evaluate the effects of low dose naltrexone compared to placebo on the activity of Crohn's disease by the following end points: Crohn's Disease Activity Index (CDAI), pain assessment, laboratory values (CRP and ESR), endoscopic appearance, histology, and quality of life surveys;
2. Examine the effects of naltrexone given over 3 months compared to 6 months for durability of response;
3. Determine the safety and toxicity of low dose naltrexone in subjects with active Crohn's disease, and
4. Study the mechanism by which naltrexone exerts its effect by measuring plasma enkephalin levels of subjects on therapy.

Purpose statement: The purpose of this study is to evaluate the effects of low dose naltrexone in a blinded placebo controlled study to determine the safety and efficacy of this compound in those with active Crohn's disease.

DETAILED DESCRIPTION:
Study design : The study is designed as a double-blind placebo controlled study for 3 months followed by a pseudo cross-over such that all subjects receiving placebo the first 3 months will receive active drug the second 3 months and all receiving naltrexone the first 3 months remain on the drug the last 3 months of this 6 month study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must give written informed consent
* Male or female subjects, > 18 years
* Patients must have endoscopic, histologic, or radiographic confirmed Crohn's Disease.
* Patients must have a Crohn's Disease Activity Index (CDAI) of at least 220 at Baseline
* Stable doses of medications for Crohn's disease over proceeding 4 weeks (for aminosalicylates and steroids: prednisone of 10mg or less daily and Entocort 3 mg/ day are allowed), and 12 weeks for azathioprine or 6-mercaptopurine.)

Exclusion Criteria:

* Subjects with ostomies or ileorectal anastomosis from prior surgical colectomy.
* Subjects who received infliximab (Remicade) within 8 weeks of study screening or humira for 4 weeks.
* Subjects requiring steroids either intravenously or prednisone >10mg /day or Entocort > 3 mg daily.
* Subjects with short-bowel syndrome.
* Abnormal liver enzymes at screening visit or known hepatitis or cirrhosis
* Hemoglobin less than 10.
* Subjects with cancer (other than skin cancer) in past 5 years.
* Women of childbearing potential unless surgically sterile or using adequate contraception (either IUD, oral or deport contraceptive, or barrier plus spermicide), and willing and able to continue contraception for 3 months after the completion of the study.
* Women who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill P. Smith, M.D., Principal Investigator — Pennsylvania State University College of Medicine
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Smith JP, Stock H, Bingaman S, Mauger D, Rogosnitzky M, Zagon IS. Low-dose naltrexone therapy improves active Crohn's disease. Am J Gastroenterol. 2007 Apr;102(4):820-8. doi: 10.1111/j.1572-0241.2007.01045.x. Epub 2007 Jan 11. PMID 17222320
- [Result] Smith JP, Bingaman SI, Ruggiero F, Mauger DT, Mukherjee A, McGovern CO, Zagon IS. Therapy with the opioid antagonist naltrexone promotes mucosal healing in active Crohn's disease: a randomized placebo-controlled trial. Dig Dis Sci. 2011 Jul;56(7):2088-97. doi: 10.1007/s10620-011-1653-7. Epub 2011 Mar 8. PMID 21380937
- See also: Penn State Hershey Clinical Trials Website — http://www.hmc.psu.edu/clinicaltrials/studies/gi/index.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, double blind, randomized placebo-controlled trial, undertaken between September 2006 and September 2009 at the Pennsylvania State University College of Medicine.
Groups:
- Placebo Then Naltrexone 4.5 mg Daily: Subjects will receive placebo for 3 months then be crossed over to active drug for an additional 3 months
- Naltrexone Then Naltrexone 4.5 mg po Daily: Group 2 will receive naltrexone 4.5 mg by mouth once a day for 6 months
Period: Overall Study
Arm/Group | Placebo Then Naltrexone 4.5 mg Daily | Naltrexone Then Naltrexone 4.5 mg po Daily
Started | 20 | 20
Completed | 19 (One patient in placebo flared and was unblinded and crossed over to active drug) | 20
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Daily: Subjects will receive placebo for 3 months then be crossed over to active drug for an additional 3 months
- Naltrexone 4.5 mg po Daily: Group 2 will receive naltrexone 4.5 mg by mouth once a day for 6 months
- Total: Total of all reporting groups
Arm/Group | Placebo Daily | Naltrexone 4.5 mg po Daily | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (2.8) | 40.5 (2.4) | 42.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Crohn's Disease Activity Index (CDAI) score [Mean (Standard Deviation); unit: CDAI score] — The CDAI score is a number unit calculated from symptoms recorded by the subject over a 7-day period before each visit, weight, hemoglobin, and physical exam findings. The score ranges from 0 to 450. A score of 220 is considered 'active' disease. A score of 150 is considered "remission." A drop of 70-points in the score is considered a "response" to therapy.
  CDAI score | 327 (19) | 365 (16) | 346 (17.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving a 70-point Decline in CDAI Scores (Crohn's Disease Activity Index) Scores;
Description: The CDAI score is a number which consists of information collected from a 7-day diary from the patient regarding symptoms. It also includes objective information from the physical exam, weight and hemotocrit. Remission is considered a score of 150 or less. Active disease is considered 220 or greater. A response to therapy is considered a decline in the CDAI score of 70-points from baseline.
Time Frame: 3 months
Measure: Number; unit: percentage of pts
Groups:
- Placebo: Placebo treated subjects for 12 weeks were analyzed for the percentage that achieved the primary outcome of a 70-point decline in the CDAI score from Baseline values
- Naltrexone 4.5 mg po Daily: Naltrexone treated subjects for 12 weeks were analyzed for the percentage that achieved the primary outcome of a 70-point decline in the CDAI score from Baseline values
Arm/Group | Placebo | Naltrexone 4.5 mg po Daily
Number analyzed (Participants) | 20 | 20
percentage of pts | 40 | 88
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 4.5 mg po Daily; The proportion of those achieving a response with a 70-point decline in CDAI score was compared between naltrexone and placebo treated subjects using the Fisher's exact test. Analysis was performed with the intent-to-treat criteria. Clinical significance was accepted if the difference met 95% confidence (p<0.05); Test type: Superiority or Other; p = 0.009, Fisher Exact — The percentage of subjects achieving a 70-point drop in CDAI score in naltrexone treated subjects was the percentage acheiving the same drop in the placebo controls

2. Secondary Outcome: Percentage Change From Baseline of Quality of Life IBDQ (Inflammatory Bowel Disease Quality of Life Survey)
Description: IBDQ (Inflammatory bowel Disease questionnaire) contains questions about health ranging from a score of poor (i.e., 32) to excellent (i.e., 224) an increase from baseline indicates improvement in quality of life.
Time Frame: Between baseline and 3 months
Population: Same as sample size calculation
Measure: Mean (Standard Error); unit: percentage of change
Groups:
- Placebo: Quality of life in subjects on placebo treatment for 12 weeks
- Naltrexone 4.5 mg po Daily: Quality of life on naltrexone treatment 12 weeks
Arm/Group | Placebo | Naltrexone 4.5 mg po Daily
Number analyzed (Participants) | 20 | 20
percentage of change | 18 (4) | 28 (5)

3. Secondary Outcome: Percentage of Patients With a 5 Point Drop in CDEIS Score by Endoscopy
Description: A secondary outcome was the appearance of the colonic mucosa on endoscopy using the Crohn's Disease Endoscopic Index of Severity (CDEIS) score described by Mary et al. Gut 1989;30:983-989.This score ranges from 0-44 based upon the extent and severity of inflammation and ulcers seen during endoscopy of the colon. A response is a drop of > 5 points from baseline. Endoscopic remission is a score of < 6 and Complete endoscopic remission is a score of > 3.
Time Frame: 12 weeks
Population: Sample size was calculated under the assumption that at least 60% of the naltrexone-treated patients, and no more than 10% of the placebo-treated patients, would respond with at least a 70-point decline in CDAI scores. With a 10% withdrawal rate, 40 subjects yields an 86% power using a two-sided, 0.05-significance level Fisher's exact test.
Measure: Number; unit: percentage of patients
Groups:
- Placebo: Placebo for 12 weeks blinded followed by naltrexone 4.5mg open labeled
- Naltrexone 4.5 mg: naltrexone 4.5 mg for 12 weeks blinded followed by naltrexone 4.5 mg open labeled
Arm/Group | Placebo | Naltrexone 4.5 mg
Number analyzed (Participants) | 20 | 20
percentage of patients | 28 [0 to 100] | 78 (.05) [0 to 100]
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 4.5 mg; Percentage of patients having a 5-point decline in the endoscopic inflammation score; Test type: Superiority or Other; p = 0.008, Fisher Exact

4. Secondary Outcome: Histology Inflammatory Score by Colon Biopsies
Description: Histology scores to assess microscopic inflammation and structural architecture were determined at baseline and after 12 weeks of either naltrexone therapy or placebo by mucosal biopsy samples obtained during colonoscopies.The pathology specimens were reviewed and scored by a Pathologist blinded to the treatment. The mean scores at baseline were the same between both groups.Differences between naltrexone and placebo treated subjects was assessed.The range in scores could be 0-25, with 0 representing no inflammation and 25 being maximum or severe inflammation..
Time Frame: 12 weeks
Population: Tissue was removed by biopsy in those undergoing colonoscopy
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Subjects who received placebo for 3 months
- Naltrexone 4.5 mg po Daily: Subjects who received naltrexone 4.5 mg by mouth once a day for 3 months
Arm/Group | Placebo | Naltrexone 4.5 mg po Daily
Number analyzed (Participants) | 20 | 20
units on a scale | 17.5 (4.5) | 5.2 (2.3)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone 4.5 mg po Daily; Test type: Superiority or Other; p = 0.048, t-test, 1 sided

ADVERSE EVENTS:
Groups:
- Placebo: Participants who received placebo for the first 12 weeks.
- Naltrexone 4.5 mg: All participants who received naltrexone either for 12 or 24 weeks.
Arm/Group | Placebo | Naltrexone 4.5 mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/40
Other Adverse Events (participants affected / at risk) | 5/20 | 5/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Naltrexone 4.5 mg (N=40)
insomnia (Nervous system disorders) | 5 (5) | 5 (5)
Fatigue (General disorders) | 3 (3) | 0 (0) — Placebo-treated subjects had increased fatigue (p = 0.04).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No